CLINICAL TRIAL: NCT05195281
Title: Pancreatic Cancer Evolution Upon Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Gabriele Capurso, Chief of Clinical Research, PancreatoBiliary Endoscopy and EUS Division, Deputy Director of Pancreas Center, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PACEUT
Record Dates: First submitted 2021-11-29; First posted 2022-01-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repetition of EUS-FNA or FNB for RNA extraction (Experimental)
  Interventions: Procedure: Fine Needle Biopsy or Aspiration

INTERVENTIONS:
Procedure: Fine Needle Biopsy or Aspiration — A new sampling of the tumor will be performed after 4-6 months of neoadjuvant chemotherapy

SUMMARY:
This project aims at evaluating the different subtypes of pancreatic cancer on EUS-tissue acquisition of pancreatic cancer patients, and their possible modifications throughout time. The study takes advantage of a systematic evaluation of pancreatic cancers through diagnostic EUS-guided fine needle biopsy (FNB) sampling of the mass performed during a restaging EUS. FNB samples represent a valuable source of cancer cells, both for the histological diagnosis and as the source of tumor macromolecules, including DNA and RNA.

Study design This is a prospective study enrolling patients with non-metastatic pancreatic cancer who already underwent diagnostic EUS with tissue acquisition and rapid on-site evaluation (ROSE) by cytologist positive for pancreatic cancer, with a first sample acquired for diagnostic purposes and a second sample stored for RNA extraction acquired with the already approved protocol BIOGASTRO.

As recommended by guidelines, patients will follow the standard pathway of treatment, being sent to chemotherapy and will then undergo restaging of the lesion and re-evaluation of vascular invasion by CT and EUS. During this second session of EUS a new specimen of the tumor will be sampled for diagnostic purposes, with a second pass undergoing for RNA extraction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing to sign informed consent
* Patient with CT scan or MRI or EUS defining the lesion as locally advanced
* Patient who already underwent EUS-TA for solid lesion of the pancreas positive for pancreatic ductal adenocarcinoma (PDAC)
* Patient undergoing neoadjuvant chemotherapy
* Patient primarily followed at San Raffaele Hospital

Exclusion Criteria:

* Patients not willing to sign informed consent
* Pregnancy and breastfeeding
* Cytology positive for malignancies other than PDAC
* Patient undergoing progression at re-staging CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2027-09-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of molecular subtype modification | 6 months
  As all patients are having baseline (at diagnosis) molecular subtype (classical or basal-like) evaluation through RNAsequencing, patients enrolled in the PACEUT trial will undergo a new evaluation of the molecular subtype (based on RNAsequencing performed on the EUS-FNA or FNB) and evaluation of gene expression

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided